CLINICAL TRIAL: NCT05773807
Title: Effect of Bispectral Index Monitoring and Observer's Assessment Alert Sedation Scale (OAA/S) Guided Sedation on Body Movement of Outpatients Undergoing Gastroscopy: a Randomized Study
Brief Title: Effect of Bispectral Index Monitoring (BIS) on Body Movement of Outpatients Undergoing Gastroscopy
Acronym: BIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-1029
Record Dates: First submitted 2023-02-20; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Gastroscopy
MeSH Terms: interventions — Consciousness Monitors; Gastroscopy; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIS group (Experimental): In the BIS group, the anesthesiologist set the TCI parameters according to the patient's height, weight, gender and age. The initial plasma target concentration was set to 1.5ug/ml, and the target concentration would be increased or decreased 0.5ug/ml every two minutes to maintain the BIS value at 45-60.
  Interventions: Other: Bispectral index; Procedure: Gastroscopy; Drug: Propofol
- OAAS/S group (Placebo Comparator): In the OAAS/S group, the anesthesiologist set the TCI parameters according to the patient's height, weight, gender and age. The initial plasma target concentration was set to 1.5ug/ml, and the target concentration would be increased or decreased 0.5ug/ml every two minutes maintain the OAA/S value at 1 point.
  Interventions: Other: Observer's assessment alert Sedation; Procedure: Gastroscopy; Drug: Propofol

INTERVENTIONS:
Other: Bispectral index — In the BIS group, the anesthesiologist set the target controlled infusion (TCI) parameters according to the patient's height, weight, gender and age. The initial plasma target concentration was set to 1.5ug/ml, and the target concentration would be increased or decreased 0.5ug/ ml every two minutes to maintain the BIS value at 45-60.
  Other Names: BIS group
  Arms: BIS group
Other: Observer's assessment alert Sedation — In the OAA/S group, the anesthesiologist set the TCI parameters according to the patient's height, weight, gender and age. The initial plasma target concentration was set to 1.5ug/ml, and the target concentration would be increased or decreased 0.5ug/ ml every two minutes maintain the OAA/S value at 1 point.
  Other Names: OAA/S group
  Arms: OAAS/S group
Procedure: Gastroscopy — Gastroscopy would be performed when the BIS value was 45-60 or the OAA/S score was 1
  Other Names: Electronic Gastroscopy
Drug: Propofol — Propofol infusion was administered under the guidance of the BIS or OAA/S before the gastroscopy, and the infusion was stopped at the end of gastroscopy
  Other Names: Propofol infusion

SUMMARY:
Patients who meet the enrollment criteria were randomized 1:1 to either the BIS group or the OAA/S group.

In the BIS group, the anesthesiologist set the target controlled infusion（TCI）parameters according to the patient's height, weight, gender and age. The initial plasma target concentration was set to 1.5 ug/ml, and the target concentration would be increased or decreased 0.5 ug/ml every two minutes to maintain the BIS value at 45-60. In the OAA/S group, the target concentration would be increased or decreased 0.5 ug/ml every two minutes to maintain the OAA/S value at 1 point.

DETAILED DESCRIPTION:
Patients who meet the enrollment criteria were randomized 1:1 to either the BIS group or the OAA/S group.

In the BIS group, the anesthesiologist set the target controlled infusion (TCI) parameters according to the patient's height, weight, gender and age. The initial plasma target concentration was set to 1.5 ug/ml, and the target concentration would be increased or decreased 0.5 ug/ml every two minutes to maintain the BIS value at 45-60. In the OAA/S group, the target concentration would be increased or decreased 0.5 ug/ml every two minutes to maintain the OAA/S value at 1 point.

Body movement, the time of gastroscopy, endoscopist satisfaction scores to sedation, the propofol consumption during gastroscopy and the time to awake were be recorded. In addition, the event of the respiration and circulation suppression during the gastroscopy were recorded. Atropine 0.3 mg was injected intravenously if bradycardia occurred (heart rate <50 beats/min), M-hydroxyamine 0.3 mg was injected intravenously if hypotension (mean arterial pressure<65 mmHg), Ephedrine 3 mg was injected if bradycardia and hypotension occured. Patients would receive face mask-assisted ventilation if the Spo2 dropped below 90% or respiratory frequency was lower than 8 breaths/min during the gastroscopy.

ELIGIBILITY:
Inclusion Criteria:

1. 18≤Age≤65 years old
2. American Society of Anaesthesiologists (ASA) Physical Status of I - II
3. 18≤BMI≤30 kg/m²
4. Outpatient patients who planned to undergo painless gastroscopy under propofol anesthesia

Exclusion Criteria:

1. Patients with communication disorders
2. Patients with alcohol and drug abuse or allergic or contraindicated drugs related to this trail
3. Patients who take anti-anxiety, depression or sedative drugs
4. Patients who participated in or were participating in other clinical trials within 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the incidence of moderate to severe body movement during gastroscopy | The time during gastroscopy, an average of 15 minutes
  Moderate to severe body movement is defined as the twisting of the patient's body due to the stimulation of the gastroscopy, making it difficult to proceed with the procedure without additional propofol.

SECONDARY OUTCOMES:
The time of gastroscopy | The time from gastroscope insertion to gastroscope withdraw, an average of 15 minutes
  The total time of gastroscopy
Endoscopist satisfaction scores | At the end of the gastroscopy
  Endoscopist satisfaction scores to sedation during gastroscopy were obtained at the end of the procedure, using a 11-point Likert scale, with 0 indicating "very dissatisfied"and 10 indicating "very satisfied"
The incidence of hypotension | The time during gastroscopy, an average of 15 minutes
  The hypotension is defined as the blood pressure<90/60 mm Hg or 20% lower at baseline
The incidence of bradycardia | The time during gastroscopy，an average of 15 minutes
  The bradycardia is defined as HR <50 beats/min
The incidence of hypoxemia | The time during gastroscopy，an average of 15 minutes
  The hypoxemia is defined as Spo2< 90%
The propofol consumption during gastroscopy | From anesthetic induction to discontinuation of propofol infusion, an average of 15 minutes
  The total propofol consumption during gastroscopy
The time to awake | The time from the end of gastroscopy to the observer's assessment alert sedation equal to 5, up to 30 minutes
  The time to awake is defined as from the end of gastroscopy to the observer's assessment alert sedation equal to 5

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, PhD, Study Chair — China, Sichuan West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No